CLINICAL TRIAL: NCT04343781
Title: National Survey of Symptoms of People Aged 70 and Overs Diagnosed With COVID-19
Acronym: COVID19PUGG2
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: ar20-0031v1
Record Dates: First submitted 2020-04-09; First posted 2020-04-13 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-04

CONDITIONS: SARS-CoV-2; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observation — observation of clinical symptoms related to COVID-19 disease

SUMMARY:
Cross-sectional study based on a French national survey aimed to described and identify the most frequent symptoms of COVID-19 older patients.

DETAILED DESCRIPTION:
This cross-sectional survey was initiated and conducted by the French Society of Geriatrics and Gerontology. A standardized questionnaire was emailed to 1600 geriatrician members of the French Society of Geriatrics and Gerontology throughout France between March 22, 2020 and April 5, 2020. Geriatricians were asked to complete the survey for their last 10 patients infected by the SARS-CoV-2. The study was declared to the Commission Nationale de l'Informatique et des Libertés (CNIL) under the number ar20-0031v1.

For each patient, demographic characteristics (age, gender, residence place, care place, autonomy according to the Groupe Iso Ressource (GIR)), medical history (presence of major neurocognitive disorder, hypertension, diabetes, asthma or chronic obstructive pulmonary disease (COPD), heart pathology, severe renal failure with a clearance of creatinine under 30ml/min, solid or liquid cancer) were collected. The symptoms within de 72 hours of the actual disease were also collected for each patient including geriatric syndromes (fall, hypoactive or hyperactive delirium, altered general status, altered conscience), general symptoms (temperature, blood pressure), respiratory symptoms (cough, polypnea), ear nose and throat (ENT) symptoms (rhinorrhea, odynophagia, otalgia, conjunctivitis, ageusia or dysgeusia, anosmia), digestive symptoms (diarrhea, nausea or vomiting), and blood formula modification (leucopenia (with count if available), lymphopenia (with count if available), thrombopenia (with count if available).

Procedure Data were collected by the physician who was in charge of the patient between March 22, 2020 and April 5, 2020.

Given the main objective of the study was only descriptive, no calculation was required concerning the number of subjects to include in the study.

ELIGIBILITY:
Inclusion Criteria:

* confirmed COVID-19 defined by a positive RT-PCR to SARS-CoV-2

Exclusion Criteria:

* none

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: all older French patients infected by SARS-CoV-2
Sampling Method: Non-Probability Sample
Enrollment: 353 (Actual)
Dates: Start 2020-03-22 (Actual); Primary Completion 2020-04-05 (Actual); Study Completion 2020-04-05 (Actual)

PRIMARY OUTCOMES:
symptoms of COVID-19 in older patients | at baseline
  description and identification of symptoms presented by older patients with confirmed COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Cédric Annweiler, M.D., Ph.D., Principal Investigator — University Hospital, Angers
Locations (1):
- Angers University Hospital, Angers, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Annweiler C, Sacco G, Salles N, Aquino JP, Gautier J, Berrut G, Guerin O, Gavazzi G. National French Survey of Coronavirus Disease (COVID-19) Symptoms in People Aged 70 and Over. Clin Infect Dis. 2021 Feb 1;72(3):490-494. doi: 10.1093/cid/ciaa792. PMID 32556328